CLINICAL TRIAL: NCT00431717
Title: Study Comparing Coronary Computed Tomography Angiography and SPECT to Detect Subclinical Coronary Atherosclerosis in Asymptomatic Diabetes
Brief Title: Coronary Computed Tomography Angiography and SPECT in Asymptomatic Diabetes
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Hyuk-Jae Chang MD, PhD, Seoul National University Bundang Hospital
Other Study IDs: B-0609/037-019
Record Dates: First submitted 2007-02-05; First posted 2007-02-06 (Estimated); Last update posted 2008-08-25 (Estimated); Status verified 2008-08

CONDITIONS: Coronary Atherosclerosis; Diabetes Mellitus
Keywords: Coronary Atherosclerosis; Diabetes Mellitus
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to compare the difference of diagnostic efficiency between coronary CT angiography and myocardial perfusion single photon emission computerized tomography in asymptomatic patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is the leading cause of death in patients with diabetes. Patients with diabetes are known to have silent myocardial ischemia more frequently than those without diabetes. Furthermore, CAD in patients with diabetes frequently manifested in advance stage, and morbidity and mortality are higher than those without diabetes. Early screening and treatment of CAD in asymptomatic patients with diabetes might reduce high morbidity and mortality.

Myocardial perfusion single photon emission computerized tomography (SPECT) is known as a gold standard method in detecting silent myocardial ischemia in asymptomatic patients with diabetes. Despite of the power of detecting myocardial ischemia functionally, there are limitations of SPECT in diagnosing subclinical coronary atherosclerosis anatomically. In recent advance in technology, coronary CT angiography (CTA) could detect subclinical coronary atherosclerosis. However, there is a paucity of information comparing the diagnostic power between SPECT and CTA.

Therefore in our study, we compare the difference of diagnostic efficiency between coronary CT angiography and myocardial perfusion single photon emission computerized tomography in asymptomatic patients with type 2 diabetes mellitus.

In this study, we will recruit asymptomatic patients with diabetes. At the time of enrollment, all patients will undergo two imaging studies (SPECT and CTA) within a few days apart. When patients had positive result in either study, they will undergo coronary angiography for confirmation. We will evaluate the results of two studies comparing with coronary angiography. When the patients are eligible for study, investigators will give information about the study and obtain written consent. The presence of chest pain symptom will be screened with Rose questionnaire. Medical history and physical examination will be performed, and baseline laboratory work-up will be performed. Investigators will evaluate the status of diabetic complication (retinopathy/nephropathy/cardiac autonomic neuropathy).

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes mellitus
2. Age 50 ~ 75 years
3. Duration of diabetes: more than 5 years
4. More than two of the following risk factors in addition to diabetes:

1)dyslipidemia, 2)hypertension, 3)smoking, 4)family history of premature coronary artery disease

Exclusion Criteria:

1. Angina pectoris or anginal equivalent symptoms
2. Insulin pump user or history of ketoacidosis
3. History of myocardial infarction, heart failure, or coronary revascularization
4. Electrocardiographic evidence of Q-wave myocardial infarction, ischemic ST- segment or T-wave changes, or complete left bundle branch block
5. Uncontrolled arrythmia
6. Hypersensitivity to contrast dye
7. Renal failure

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Asymptomtaic type 2 diabetes mellitus with multiple risk factors
Sampling Method: Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2006-11; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Huk-Jae Chang, MD, PhD, Study Director — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang hospital, Sungnam-si, Gyeonggi-do, South Korea